CLINICAL TRIAL: NCT02383238
Title: Randomized, Placebo Controlled, Crossover Clinical Study to Analyse the Effect of Dapagliflozin on Microvascular and Macrovascular Circulation and Total Body Sodium Content
Brief Title: Effect of Dapagliflozin on Microvascular and Macrovascular Circulation and Total Body Sodium Content
Acronym: Dapa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Roland E. Schmieder, Prof. Dr. Roland E. Schmieder, University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MB102-210
Record Dates: First submitted 2014-07-24; First posted 2015-03-09 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Dapagliflozin; diabetes mellitus; vascular
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dapagliflozin (Active Comparator): Dapagliflozin, 10 mg/day, oral administration, 6 weeks
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo, oral administration, 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg, oral for 6 weeks
  Other Names: Forxiga
  Arms: Dapagliflozin
Drug: Placebo — oral for 6 weeks
  Arms: Placebo

SUMMARY:
Dapagliflozin leads to improved vascular function in the micro- and macrocirculation by action on various cardiovascular risk factors, in particular by effectively controlling hyperglycemia, arterial hypertension and reducing whole sodium content amongst others.

DETAILED DESCRIPTION:
Diabetes mellitus, considered at the beginning as a metabolic disorder, mutates into a predominantly vascular disease, once its duration extends over several years or/and when additional cardiovascular risk factors coexist, in particular arterial hypertension. In accordance, patients with type 2 diabetes die because of microvascular and macrovascular complications, and only rarely because of hypoglycaemic or hyperglycaemic shock syndromes [1]. As a consequence, treatment of type 2 diabetes should focus not only on metabolic control but also on improving the global vascular risk. Analyses that have compared the importance of the various cardiovascular risk factors concluded that reductions of blood pressure and lipid levels are significantly more important than reduction of hyperglycemia [2]. Of course, a multidisciplinary approach is desirable and the STENO-2 study has clearly indicated that in mid-term microvascular complications and in long-term macrovascular complications can be prevented in type 2 diabetes [3].

Vascular changes occurring in the course of type 2 diabetes, arterial hypertension and elevated global cardiovascular risk can now reliably assessed non-invasively, and already at the very early stage of vascular remodeling processes. For example, the guidelines of the European Society of Hypertension recommend several vascular

#0284 CSP 130911 v1.4.docx 8 parameters to be assessed already at the diagnosis of the disease in order to analyze early organ damage of the arteries [4]. The measurement of pulse wave velocity, pulse wave analysis, central (aortic) systolic pressure and pulse pressure are tools to detect early vascular changes in the large arteries related to a faster wave reflection in the arterial tree [5]. Wall to lumen ratio of retinal arteries, retinal capillary flow and flow mediated vasodilation are tools to detect changes in the microvascular circulation [6]. These parameters are only infrequently measured in studies with type 2 diabetes, mainly due to lack of awareness that the vascular changes are the key prognostic factor in type-2 diabetes that ultimately determine the fate of the patient.

Dapagliflozin is a novel selective SLGT-2 inhibitor that has been shown to improve glycaemic control after 2, 12, and 24 weeks as well as after 1 and 2 years. Dapagliflozin produced dose dependent increases in glucosuria and clinically meaningful changes of glycemic parameters in type 2 diabetes in addition to weight loss. Most striking, dapagliflozin was also found to lower systolic blood pressure by 5 mmHg. This reduction in blood pressure might be related to weight loss or/and concomitant loss of total body sodium content. However, the precise mechanism of the blood pressure reduction needs to be elucidated. Loss of sodium would lead to a less reactive contraction of the small arteries in response to increased sympathetic activity, angiotensin II [7] and catecholamines.

In summary, dapagliflozin exert beneficial effects on a variety of cardiovascular risk factors, such as hyperglycaemia, hypertension and obesity. These changes should lead (so the hypothesis) to improved vascular function in the micro- and macrocirculation. Moreover, increased total body content of sodium that now can be measured in humans by a specific MRI technique [8] may also be reduced by dapagliflozin that may lead to less vasoreactive responses since the tubular SGLT-2 mediated glucose uptake is sodium related, i.e. blockade should lead to sodium loss. However, the latter is nothing more than hypothesis and requires clear proof by clinical studies in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. HbA1c > 6.5%
3. age > 18 years
4. male and females

Exclusion Criteria:

1. age > 75 years
2. HbA1c > 10 %,
3. reduced renal function (eGFR < 60 ml/min/1.73 m²).
4. insulin therapy, or any antidiabetic medication other than metformin.
5. uncontrolled hypertension (> 180/>110 mmHg)
6. cardiovascular event within the last 3 months
7. Use of loop diuretics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Microcirculation | 6 weeks
  To analyse the effects after 6 weeks of treatment with dapagliflozin on retinal capillary flow (given as AU) as the key measurement of vascular remodeling in the microcirculation compared to placebo.

SECONDARY OUTCOMES:
Macrovascular circulation | 6 weeks
  To analyse the effects after 6 weeks of treatment with dapagliflozin on central (aortic) systolic pressure, central (aortic) pulse pressure and augmentation pressure, on retinal capillary flow after flicker light exposure, parameters that all are determined by pulse wave reflection (i.e. arterial wall properties) in the arterial tree compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Schmieder, Prof., Principal Investigator — Department of Medicine 4, University of Erlangen-Nuernberg
Locations (1):
- University Erlangen-Nuernberg, Erlangen, Germany

REFERENCES:
- [Result] Karg MV, Bosch A, Kannenkeril D, Striepe K, Ott C, Schneider MP, Boemke-Zelch F, Linz P, Nagel AM, Titze J, Uder M, Schmieder RE. SGLT-2-inhibition with dapagliflozin reduces tissue sodium content: a randomised controlled trial. Cardiovasc Diabetol. 2018 Jan 4;17(1):5. doi: 10.1186/s12933-017-0654-z. PMID 29301520
- [Derived] Staef M, Ott C, Kannenkeril D, Striepe K, Schiffer M, Schmieder RE, Bosch A. Determinants of arterial stiffness in patients with type 2 diabetes mellitus: a cross sectional analysis. Sci Rep. 2023 Jun 2;13(1):8944. doi: 10.1038/s41598-023-35589-4. PMID 37268640
- [Derived] Gessner A, Gemeinhardt A, Bosch A, Kannenkeril D, Staerk C, Mayr A, Fromm MF, Schmieder RE, Maas R. Effects of treatment with SGLT-2 inhibitors on arginine-related cardiovascular and renal biomarkers. Cardiovasc Diabetol. 2022 Jan 6;21(1):4. doi: 10.1186/s12933-021-01436-x. PMID 34991562
- [Derived] Kannenkeril D, Jung S, Harazny J, Striepe K, Ott C, Dahlmann A, Kopp C, Schiffer M, Linz P, Nagel AM, Uder M, Schmieder RE. Tissue sodium content correlates with hypertrophic vascular remodeling in type 2 diabetes. J Diabetes Complications. 2021 Dec;35(12):108055. doi: 10.1016/j.jdiacomp.2021.108055. Epub 2021 Sep 29. PMID 34620556
- [Derived] Kannenkeril D, Bosch A, Harazny J, Karg M, Jung S, Ott C, Schmieder RE. Early vascular parameters in the micro- and macrocirculation in type 2 diabetes. Cardiovasc Diabetol. 2018 Sep 19;17(1):128. doi: 10.1186/s12933-018-0770-4. PMID 30231923
- [Derived] Ott C, Jumar A, Striepe K, Friedrich S, Karg MV, Bramlage P, Schmieder RE. A randomised study of the impact of the SGLT2 inhibitor dapagliflozin on microvascular and macrovascular circulation. Cardiovasc Diabetol. 2017 Feb 23;16(1):26. doi: 10.1186/s12933-017-0510-1. PMID 28231831